CLINICAL TRIAL: NCT03144427
Title: The Acute Burn Resuscitation Multicenter Prospective Observational Trial
Acronym: ABRUPT
Status: Completed | Type: Observational
Sponsor: American Burn Association (Other)
Collaborators: U.S. Army Medical Research Acquisition Activity (U.S. Federal Agency); University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: ABuRN-001; W81XWH-16-2-0048 Log#MB150076 (Other Grant/Funding Number: U.S. Army Medical Research Acquisition Activity)
Record Dates: First submitted 2017-04-27; First posted 2017-05-08 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Burns; Shock
Keywords: albumin; resuscitation; burns; shock; fluid creep
MeSH Terms: conditions — Burns; Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Burns: Patients with burns to 20% or more of their BSA (body surface area) require resuscitation with intravenous crystalloid fluids in order to avoid organ failure and death

SUMMARY:
This is a prospective, non-interventional, observational study of consecutive burn patients admitted to 20 selected burn centers in North America. Primarily, data collection will be continuous "real-time" documentation of fluid infusion rates, vital signs and laboratory values of patients receiving fluid resuscitation during the first 48 hours following burn injury. All aspects of the resuscitation and all investigations performed will be according to the participating center's regular protocol, as this is purely an observational and non-interventional study. Further data collection on outcomes (organ function, ventilation duration, length of stay, and survival) will be collected at 72h, 96 h, and at hospital discharge.

DETAILED DESCRIPTION:
This is a prospective observational study with no intervention. Study sites have been selected to include wide cross-representation of resuscitation practices using crystalloids alone, crystalloid plus albumin, and among sites that use albumin, variable approaches to the timing of albumin initiation.

Detailed data will be continuously collected in "real time" during fluid resuscitation over the 1st 48 hours following a burn injury. Data collection during this phase will be done prospectively, hour-by-hour, by the bedside nurse caring for the patient. Primarily this data collection will involve recording of resuscitation fluid volumes, urinary output, vital signs (heart rate and blood pressure), and use of vasopressors and inotropes. Outcome data (organ function, need for mechanical ventilation, hospital length of stay, and survival) will be collected at various time points during the subjects' acute care stay.

At completion of the study we intend to make the following comparisons:

1. Subjects that received crystalloids only compared to subjects that received crystalloids plus albumin.
2. Subjects that had albumin started "early" (< 8 hours post burn), compared to subjects that had albumin started "intermediate" (8-12 hours post burn), compared to subjects that had albumin started "late" (>12 hours post burn).
3. Characteristics of resuscitation prior to the start of albumin ("pre-albumin") compared to characteristics of resuscitation following initiation of albumin ("post albumin").

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* ≥ 20% TBSA burns
* Admitted to the burn center ≤ 12 post injury

Exclusion Criteria:

* Significant associated trauma
* High voltage (≥ 1000 volts) electrical burns
* Surgery anticipated within 48 hours from injury
* Fresh frozen plasma (FFP) anticipated to be given at any time ≤ 48 hours from injury
* Hypertonic saline (HTS) anticipated to be given at any time ≤ 48 hours from injury
* Hydroxyethyl starch (HES) anticipated to be given at any time ≤ 48 hours from injury
* High dose Vitamin C infusion is anticipated to be given at any time ≤ 48 hours from injury
* Death occurs or comfort measures are instituted within ≤ 48 hours from injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients must be ≥ 18 years of age with a TBSA burn of ≥ 20%, and they must have been admitted to the burn center ≤ 12 hours following the injury.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2017-02-24 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Fluid resuscitation volume | 24 hours post burn injury
  Total fluid resuscitation volume in mL/kg/% TBSA (total body surface area) burn
albumin : crystalloid ratio | 24 hours hours post burn injury
  albumin : crystalloid ratio ( mL albumin : mL crystalloid, and, grams albumin : mL crystalloid)
Fluid resuscitation volume | 48 hours post burn injury
  Total fluid resuscitation volume in mL/kg/% TBSA burn
albumin : crystalloid ratio | 48 hours post burn injury
  albumin : crystalloid ratio ( mL albumin : mL crystalloid, and, grams albumin : mL crystalloid)

SECONDARY OUTCOMES:
I/O Ratio | 24 hours post burn injury
  Total intake and output ratio
I/O Ratio | 48 hours post burn injury
  Total intake and output ratio
Doses of vasopressors and inotropes | 24 hours post burn injury
  Total doses of vasopressors and inotropes
Doses of vasopressors and inotropes | 48 hours post burn injury
  Total doses of vasopressors and inotropes
Fasciotomy | during the first 48 hours post burn injury
  Documentation of fasciotomy performed
abdominal compartment syndrome | during the first 48 hours post burn injury
  Occurrence of abdominal compartment syndrome
completion of resuscitation | up to 48 hours post burn injury
  Time to completion of resuscitation
AKIN Score (acute kidney injury network) | 24 hours post burn injury
  Acute Kidney Injury Network stage
AKIN Score | 48 hours post burn injury
  Acute Kidney Injury Network stage
AKIN Score | 72 hours post burn injury
  Acute Kidney Injury Network stage
AKIN Score | 96 hours post burn injury
  Acute Kidney Injury Network stage
SOFA score (sequential organ failure assessment) | 24 hours post burn injury
  Sequential Organ Failure Assessment
SOFA score | 48 hours post burn injury
  Sequential Organ Failure Assessment
SOFA score | 72 hours post burn injury
  Sequential Organ Failure Assessment
SOFA score | 96 hours post burn injury
  Sequential Organ Failure Assessment
Mechanical Ventilation | from date of hospital admit until date of hospital discharge, assessed over duration of hospitalization up to 12 months
  Duration of mechanical ventilation and ventilator free days
Hospital Stay | from date of hospital admit until date of hospital discharge, assessed over duration of hospitalization up to 12 months
  Length of hospital stay
Survival | 28 days post burn injury or death, whichever occurs first
  In hospital and 28 day survival

CONTACTS AND LOCATIONS:
Overall Officials: David Greenhalgh, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Medical Center-Regional Burn Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pruitt BA Jr. Protection from excessive resuscitation: "pushing the pendulum back". J Trauma. 2000 Sep;49(3):567-8. doi: 10.1097/00005373-200009000-00030. No abstract available. PMID 11003341
- [Background] Zak AL, Harrington DT, Barillo DJ, Lawlor DF, Shirani KZ, Goodwin CW. Acute respiratory failure that complicates the resuscitation of pediatric patients with scald injuries. J Burn Care Rehabil. 1999 Sep-Oct;20(5):391-9. doi: 10.1097/00004630-199909000-00011. PMID 10501327
- [Background] Hobson KG, Young KM, Ciraulo A, Palmieri TL, Greenhalgh DG. Release of abdominal compartment syndrome improves survival in patients with burn injury. J Trauma. 2002 Dec;53(6):1129-33; discussion 1133-4. doi: 10.1097/00005373-200212000-00016. PMID 12478039
- [Background] Klein MB, Hayden D, Elson C, Nathens AB, Gamelli RL, Gibran NS, Herndon DN, Arnoldo B, Silver G, Schoenfeld D, Tompkins RG. The association between fluid administration and outcome following major burn: a multicenter study. Ann Surg. 2007 Apr;245(4):622-8. doi: 10.1097/01.sla.0000252572.50684.49. PMID 17414612
- [Background] Holcomb JB, del Junco DJ, Fox EE, Wade CE, Cohen MJ, Schreiber MA, Alarcon LH, Bai Y, Brasel KJ, Bulger EM, Cotton BA, Matijevic N, Muskat P, Myers JG, Phelan HA, White CE, Zhang J, Rahbar MH; PROMMTT Study Group. The prospective, observational, multicenter, major trauma transfusion (PROMMTT) study: comparative effectiveness of a time-varying treatment with competing risks. JAMA Surg. 2013 Feb;148(2):127-36. doi: 10.1001/2013.jamasurg.387. PMID 23560283
- [Background] Holcomb JB, Fox EE, Wade CE; PROMMTT Study Group. The PRospective Observational Multicenter Major Trauma Transfusion (PROMMTT) study. J Trauma Acute Care Surg. 2013 Jul;75(1 Suppl 1):S1-2. doi: 10.1097/TA.0b013e3182983876. No abstract available. PMID 23778505
- [Background] Rahbar MH, Fox EE, del Junco DJ, Cotton BA, Podbielski JM, Matijevic N, Cohen MJ, Schreiber MA, Zhang J, Mirhaji P, Duran SJ, Reynolds RJ, Benjamin-Garner R, Holcomb JB; PROMMTT Investigators. Coordination and management of multicenter clinical studies in trauma: Experience from the PRospective Observational Multicenter Major Trauma Transfusion (PROMMTT) Study. Resuscitation. 2012 Apr;83(4):459-64. doi: 10.1016/j.resuscitation.2011.09.019. Epub 2011 Oct 12. PMID 22001613
- [Background] Holcomb JB, Tilley BC, Baraniuk S, Fox EE, Wade CE, Podbielski JM, del Junco DJ, Brasel KJ, Bulger EM, Callcut RA, Cohen MJ, Cotton BA, Fabian TC, Inaba K, Kerby JD, Muskat P, O'Keeffe T, Rizoli S, Robinson BR, Scalea TM, Schreiber MA, Stein DM, Weinberg JA, Callum JL, Hess JR, Matijevic N, Miller CN, Pittet JF, Hoyt DB, Pearson GD, Leroux B, van Belle G; PROPPR Study Group. Transfusion of plasma, platelets, and red blood cells in a 1:1:1 vs a 1:1:2 ratio and mortality in patients with severe trauma: the PROPPR randomized clinical trial. JAMA. 2015 Feb 3;313(5):471-82. doi: 10.1001/jama.2015.12. PMID 25647203
- [Background] Cartotto R, Callum J. A review of the use of human albumin in burn patients. J Burn Care Res. 2012 Nov-Dec;33(6):702-17. doi: 10.1097/BCR.0b013e31825b1cf6. PMID 23143614
- [Background] Baxter CR, Shires T. Physiological response to crystalloid resuscitation of severe burns. Ann N Y Acad Sci. 1968 Aug 14;150(3):874-94. doi: 10.1111/j.1749-6632.1968.tb14738.x. No abstract available. PMID 4973463
- [Background] Baxter CR, Marvin J, Curreri PW. Fluid and electrolyte therapy of burn shock. Heart Lung. 1973 Sep-Oct;2(5):707-13. No abstract available. PMID 4490375
- [Background] Pruitt BA Jr. Fluid and electrolyte replacement in the burned patient. Surg Clin North Am. 1978 Dec;58(6):1291-1312. doi: 10.1016/s0039-6109(16)41692-0. No abstract available. PMID 734610
- [Background] Pruitt BA Jr. The burn patient: II. Later care and complications of thermal injury. Curr Probl Surg. 1979 May;16(5):1-95. doi: 10.1016/s0011-3840(79)80009-x. PMID 376227
- [Background] Cartotto RC, Innes M, Musgrave MA, Gomez M, Cooper AB. How well does the Parkland formula estimate actual fluid resuscitation volumes? J Burn Care Rehabil. 2002 Jul-Aug;23(4):258-65. doi: 10.1097/00004630-200207000-00006. PMID 12142578
- [Background] Engrav LH, Colescott PL, Kemalyan N, Heimbach DM, Gibran NS, Solem LD, Dimick AR, Gamelli RL, Lentz CW. A biopsy of the use of the Baxter formula to resuscitate burns or do we do it like Charlie did it? J Burn Care Rehabil. 2000 Mar-Apr;21(2):91-5. doi: 10.1097/00004630-200021020-00002. PMID 10752739
- [Background] Cancio LC, Chavez S, Alvarado-Ortega M, Barillo DJ, Walker SC, McManus AT, Goodwin CW. Predicting increased fluid requirements during the resuscitation of thermally injured patients. J Trauma. 2004 Feb;56(2):404-13; discussion 413-4. doi: 10.1097/01.TA.0000075341.43956.E4. PMID 14960986
- [Background] Cartotto R, Zhou A. Fluid creep: the pendulum hasn't swung back yet! J Burn Care Res. 2010 Jul-Aug;31(4):551-8. doi: 10.1097/BCR.0b013e3181e4d732. PMID 20616649
- [Background] Saffle JI. The phenomenon of "fluid creep" in acute burn resuscitation. J Burn Care Res. 2007 May-Jun;28(3):382-95. doi: 10.1097/BCR.0B013E318053D3A1. PMID 17438489
- [Background] Recinos PR, Hartford CA, Ziffren SE. Fluid resuscitation of burn patients comparing a crystalloid with a colloid containing solution: a prospective study. J Iowa Med Soc. 1975 Oct;65(10):426-32. No abstract available. PMID 1194720
- [Background] Jelenko C 3rd, Williams JB, Wheeler ML, Callaway BD, Fackler VK, Albers CA, Barger AA. Studies in shock and resuscitation, I: use of a hypertonic, albumin-containing, fluid demand regimen (HALFD) in resuscitation. Crit Care Med. 1979 Apr;7(4):157-67. PMID 446052
- [Background] Goodwin CW, Dorethy J, Lam V, Pruitt BA Jr. Randomized trial of efficacy of crystalloid and colloid resuscitation on hemodynamic response and lung water following thermal injury. Ann Surg. 1983 May;197(5):520-31. doi: 10.1097/00000658-198305000-00004. PMID 6342554
- [Background] Cooper AB, Cohn SM, Zhang HS, Hanna K, Stewart TE, Slutsky AS; ALBUR Investigators. Five percent albumin for adult burn shock resuscitation: lack of effect on daily multiple organ dysfunction score. Transfusion. 2006 Jan;46(1):80-9. doi: 10.1111/j.1537-2995.2005.00667.x. PMID 16398734
- [Background] Lawrence A, Faraklas I, Watkins H, Allen A, Cochran A, Morris S, Saffle J. Colloid administration normalizes resuscitation ratio and ameliorates "fluid creep". J Burn Care Res. 2010 Jan-Feb;31(1):40-7. doi: 10.1097/BCR.0b013e3181cb8c72. PMID 20061836
- [Background] Faraklas I, Lam U, Cochran A, Stoddard G, Saffle J. Colloid normalizes resuscitation ratio in pediatric burns. J Burn Care Res. 2011 Jan-Feb;32(1):91-7. doi: 10.1097/BCR.0b013e318204b379. PMID 21131844
- [Background] 25. Mehrkens HH, Ahnefeld FW. Volume and fluid replacement in the early post burn period: an animal experimental study. Burns 1979;5:113-15
- [Background] Asch MJ, Feldman RJ, Walker HL, Foley FD, Popp RL, Mason AD Jr, Pruitt BA Jr. Systemic and pulmonary hemodynamic changes accompanying thermal injury. Ann Surg. 1973 Aug;178(2):218-21. doi: 10.1097/00000658-197308000-00020. No abstract available. PMID 4723430
- [Background] Demling RH, Kramer G, Harms B. Role of thermal injury-induced hypoproteinemia on fluid flux and protein permeability in burned and nonburned tissue. Surgery. 1984 Feb;95(2):136-44. PMID 6695330
- [Background] Demling RH, Kramer GC, Gunther R, Nerlich M. Effect of nonprotein colloid on postburn edema formation in soft tissues and lung. Surgery. 1984 May;95(5):593-602. PMID 6200946
- [Background] Onarheim H, Reed RK. Thermal skin injury: effect of fluid therapy on the transcapillary colloid osmotic gradient. J Surg Res. 1991 Mar;50(3):272-8. doi: 10.1016/0022-4804(91)90190-w. PMID 1999916
- [Background] Moncrief JA. Effect of various fluid regimens and pharmacologic agents on the circulatory hemodynamics of the immediate postburn period. Ann Surg. 1966 Oct;164(4):723-52. doi: 10.1097/00000658-196610000-00017. No abstract available. PMID 5924792
- [Background] Park SH, Hemmila MR, Wahl WL. Early albumin use improves mortality in difficult to resuscitate burn patients. J Trauma Acute Care Surg. 2012 Nov;73(5):1294-7. doi: 10.1097/TA.0b013e31827019b1. PMID 23117385